CLINICAL TRIAL: NCT03650426
Title: Comparison Between the Onlay and Inlay Techniques for Patellar Resurfacing in Posterior Cruciate Ligament-Substituting Total Knee Arthroplasty: A Prospective, Randomized Controlled Trial
Brief Title: Comparison Between the Onlay and Inlay Techniques for Patellar Resurfacing in Posterior Cruciate Ligament-Substituting Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COA 017/2561
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2018-07

CONDITIONS: Onlay Patellar Resurfacing Technique; Inlay Patellar Resurfacing Technique; Patellar Resurfacing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Onlay patellar resurfacing technique (Active Comparator)
  Interventions: Procedure: Total knee with onlay patellar resurfacing technique
- Inlay patellar resurfacing technique (Experimental)
  Interventions: Procedure: Total knee with inlay patellar resurfacing technique

INTERVENTIONS:
Procedure: Total knee with onlay patellar resurfacing technique — The patellar resurfacing technique that the patellar implant is embedded on the patellar bone.The patellar implant is placed on top of a flat tibial osteotomy or cut-surfaced bone
  Arms: Onlay patellar resurfacing technique
Procedure: Total knee with inlay patellar resurfacing technique — The patellar resurfacing technique that the patellar implant is embedded in the patellar bone.The patellar implant is surrounded by a rim of cortical bone and supported by hardened, sclerotic bone
  Arms: Inlay patellar resurfacing technique

SUMMARY:
The purpose of this study is to compare clinical outcome in posterior cruciate ligament-substituting total knee arthroplasty with onlay patellar resurfacing technique and inlay patellar resurfacing technique

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of knee who were scheduled for a primary total knee arthroplasty

Exclusion Criteria:

* Valgus deformity
* History of inflammatory arthroplathy
* Previous fracture or open surgery on the same knee
* History of patellar instability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Change of post-operative anterior knee pain | Change from baseline Visual Analog Scale for anterior knee pain at 3 months, 6 months, and 12 months after surgery
  Visual Analog Scale for anterior knee pain (minimum 0, maximum 10) Do higher values represent a worse outcome
range of motion of knee | Change from baseline Knee Society and Knee Society function score at 3 months, 6 months, and 12 months after surgery
  Knee Society and Knee Society function score (minimum 0, maximum 200)
Knee Society and Knee Society function score | Change from baseline Knee Society and Knee Society function score at 3 months, 6 months, and 12 months after surgery
  Knee Society and Knee Society function score (minimum 0, maximum 200)
New patellar score | Change from baseline new patellar score at 3 months, 6 months, and 12 months after surgery
  New patellar score (minimum 0, maximum 30)
Oxford knee score | Change from baseline Oxford knee score 3 months, 6 months, and 12 months after surgery
  Oxford knee score (minimum 0, maximum 48)
Prevalence of anterior knee pain ,AKP | Change from baseline Prevalence of anterior knee pain ,AKP 3 months, 6 months, and 12 months after surgery
  Prevalence of anterior knee pain ,AKP (minimum 0, maximum 10)
Prevalence of patellar crepitus complication | Change from baseline patellar crepitus complication 3 months, 6 months, and 12 months after surgery
  Prevalence of patellar crepitus complication (present, absent)

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — Department of Orthopaedics, Faculty of Medicine Vajira Hospital, Navamindradhiraj University
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand